CLINICAL TRIAL: NCT00662792
Title: A Randomised, Double-blind Clinical Efficacy and Safety Comparison of Tiotropium/Salmeterol 7.5/25 Inhalation Powder in the Morning Via Tiotropium/Salmeterol HandiHaler, Tiotropium 18 Mcg Inhalation Powder in the Morning Via Spiriva HandiHaler, Salmeterol 50 Mcg MDPI in the Morning and Evening and the Free Combination Tiotropium 18 Mcg Inhalation Powder in the Morning Via Spiriva HandiHaler Plus Salmeterol 50 Mcg MDPI in the Morning and Evening Following Chronic Administration (6-week Treatment Periods) in Patients With COPD
Brief Title: Efficacy and Safety Comparison of Tiotropium Daily + Salmeterol Daily or Twice Daily Versus Tiotropium Daily in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1184.13
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- T+S_PE/ Tio18GEL / Salm50DPI / T18GEL+S_DPI (Experimental): 7.5 µg/ 25 µg Tiotropium/Salmeterol (T+S_PE)/ 18 µg Tiotropium (Tio18GEL) / 50 µg Salmeterol MDPI (Salm50DPI) / 18 µg Tiotropium (T18GEL) plus 50 µg Salmeterol MDPI (S_DPI) BID
  Interventions: Drug: Tiotropium (Tio18GEL); Drug: Salmeterol MDPI (Salm50DPI); Drug: Tiotropium (T18GEL) + Salmeterol MDPI (S_DPI); Drug: Tiotropium/Salmeterol (T+S_PE)
- Tio18GEL/ T18GEL+S_DPI/ T+S_PE/ Salm50DPI (Experimental): 18 µg Tiotropium (Tio18GEL) / 18 µg Tiotropium (T18GEL) + 50 µg Salmeterol MDPI (S_DPI) BID / 7.5 µg/ 25 µg Tiotropium/Salmeterol (T+S_PE) / 50 µg Salmeterol MDPI (Salm50DPI)
  Interventions: Drug: Tiotropium (Tio18GEL); Drug: Salmeterol MDPI (Salm50DPI); Drug: Tiotropium (T18GEL) + Salmeterol MDPI (S_DPI); Drug: Tiotropium/Salmeterol (T+S_PE)
- Salm50DPI/ T+S_PE/ T18GEL+S_DPI/ Tio18GEL (Experimental): 50 µg Salmeterol MDPI (Salm50DPI) / 7.5 µg/ 25 µg Tiotropium/Salmeterol (T+S_PE) / 18 µg Tiotropium (T18GEL) + 50 µg Salmeterol MDPI (S_DPI) BID / 18 µg Tiotropium (Tio18GEL)
  Interventions: Drug: Tiotropium (Tio18GEL); Drug: Salmeterol MDPI (Salm50DPI); Drug: Tiotropium (T18GEL) + Salmeterol MDPI (S_DPI); Drug: Tiotropium/Salmeterol (T+S_PE)
- T18GEL+S_DPI/ Salm50DPI/ Tio18GEL/ T+S_PE (Experimental): 18 µg Tiotropium (T18GEL) + 50 µg Salmeterol MDPI (S_DPI) BID / 50 µg Salmeterol MDPI (Salm50DPI) / 18 µg Tiotropium (Tio18GEL) / 7.5 µg/ 25 µg Tiotropium/Salmeterol (T+S_PE)
  Interventions: Drug: Tiotropium (Tio18GEL); Drug: Salmeterol MDPI (Salm50DPI); Drug: Tiotropium (T18GEL) + Salmeterol MDPI (S_DPI); Drug: Tiotropium/Salmeterol (T+S_PE)

INTERVENTIONS:
Drug: Tiotropium (Tio18GEL) — 18 µg Tiotropium (Tio18GEL) inhalation powder
Drug: Salmeterol MDPI (Salm50DPI) — 50 µg Salmeterol MDPI (Salm50DPI) twice daily (BID)
Drug: Tiotropium (T18GEL) + Salmeterol MDPI (S_DPI) — 18 µg Tiotropium (T18GEL) inhalation powder plus 50 µg Salmeterol MDPI (S_DPI) twice daily (BID)
Drug: Tiotropium/Salmeterol (T+S_PE) — Fixed-dose combination of 7.5 µg/ 25 µg Tiotropium/Salmeterol (T+S_PE) inhalation powder

SUMMARY:
The primary objective of this trial is to establish superiority of the once-daily Tiotropium plus Salmeterol Inhalation Powder in daytime lung function response and non-inferiority in night-time lung function response over the comparator treatments inhaled in their established dose regimens when administered for 6-week periods to patients with chronic obstructive pulmonary disease (COPD). The main secondary objective is to evaluate the safety of the Tiotropium plus Salmeterol Inhalation Powder versus the comparator treatments.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with ICH-GCP guidelines and local legislations prior to any study-related procedures, which includes medication washout and restrictions.
2. All patients must have a diagnosis of COPD and must meet the following criteria:

   relatively stable* airway obstruction with a post-bronchodilator FEV1 < 80% of predicted normal and post-bronchodilator FEV1 < 70% of post-bronchodilator FVC at Visit 1 (according to GOLD criteria).

   * The randomisation of patients with any respiratory infection or COPD exacerbation in the 6 weeks prior to the Screening Visit (Visit 1) or during the baseline period should be postponed. Patients may be randomised 6 weeks following recovery from the infection or exacerbation. Predicted normal values will be calculated according to ECSC.
3. Male or female patients 40 years of age or older.
4. Patients must be current or ex-smokers with a smoking history of 10 pack-years.
5. Patients must be able to perform technically acceptable pulmonary function tests
6. Patients must be able to inhale medication in a competent manner.
7. Patients must be able to perform all necessary recordings in the diary.

Exclusion Criteria:

1. Significant diseases other than COPD
2. Patients with clinically significant abnormal baseline haematology, blood chemistry or urinalysis, if the abnormality defines a significant disease as defined in exclusion criterion No. 1.
3. Patients with a recent history of myocardial infarction.
4. Patients with any unstable or life-threatening cardiac arrhythmia requiring intervention or change in drug therapy during the past year.
5. Hospitalisation for cardiac failure during the past year.
6. Malignancy within the last five years excluded basal cell carcinoma.
7. Patients with a history of asthma or who have a total blood eosinophil count 600/mm3.
8. Patients with a history of life threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis.
9. Known active tuberculosis.
10. Patients with a history of alcohol or drug abuse.
11. Thoracotomy with pulmonary resection.
12. Rehabilitation program within the last six weeks
13. Patients who regularly use daytime oxygen therapy
14. Patients who have taken an investigational drug within 30 days
15. Use of not allowed medications
16. Known hypersensitivity to used drugs or other components of the study medication.
17. Pregnant or nursing women
18. Women of childbearing potential not using a highly effective method of birth control. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner. Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.
19. Patients who are currently participating in another study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2008-04-15 (Actual); Primary Completion 2009-07-22 (Actual); Study Completion 2009-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- Germany (12):
  - 1184.13.1302 Boehringer Ingelheim Investigational Site, Berlin
  - 1184.13.1309 Boehringer Ingelheim Investigational Site, Berlin
  - 1184.13.1308 Boehringer Ingelheim Investigational Site, Cottbus
  - 1184.13.1311 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1184.13.1312 Boehringer Ingelheim Investigational Site, Hamburg
  - 1184.13.1305 Boehringer Ingelheim Investigational Site, Mainz
  - 1184.13.1301 Boehringer Ingelheim Investigational Site, Mannheim
  - 1184.13.1306 Boehringer Ingelheim Investigational Site, Rodgau-Dudenhofen
  - 1184.13.1310 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1184.13.1307 Boehringer Ingelheim Investigational Site, Schwerin
  - 1184.13.1304 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 1184.13.1303 Boehringer Ingelheim Investigational Site, Wiesloch

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised, double-blind, 4-way crossover efficacy and safety comparison of Tiotropium/Salmeterol, Tiotropium Salmeterol and the free combination Tiotropium plus Salmeterol (50 μg) following chronic Administration in patients with COPD.
  Patients received each of the 4 treatments for 6 weeks in a randomised sequence.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- T+S_PE/ Tio18GEL / Salm50DPI / T18GEL+S_DPI: Period 1: Fixed-dose combination of 7.5 µg/ 25 µg Tiotropium/Salmeterol (T+S_PE) inhalation powder from one capsule via the blue HandiHaler® once daily (QD) in the morning, one capsule of matching placebo via the grey HandiHaler® and one actuation from the placebo Multi-Dose Powder Inhaler (MDPI) in the morning and one actuation from the placebo MDPI in the evening.
  Period 2: 18 µg Tiotropium (Tio18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® QD in the morning, one capsule of matching placebo via the blue HandiHaler® and one actuation from the placebo MDPI in the morning and one actuation from the placebo MDPI in the evening.
  Period 3: One actuation of 50 µg Salmeterol MDPI (Salm50DPI) twice daily (BID), in the morning and in the evening, one capsule of matching placebo from grey HandiHaler® and one capsule of matching placebo from the blue HandiHaler® in the morning.
  Period 4: 18 µg Tiotropium (T18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® in the morning plus one actuation of 50 µg Salmeterol MDPI (S_DPI) BID, in the morning and in the evening, and one placebo capsule from blue Handi Haler® in the morning.
  Each dose of study medication had to be taken approximately at the same time, with 12 hours between the evening and morning dose. Each treatment period was 6 weeks on average with no wash-out between the treatment periods.
- Tio18GEL/ T18GEL+S_DPI/ T+S_PE/ Salm50DPI: Period 1: 18 µg Tiotropium (Tio18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® QD in the morning, one capsule of matching placebo via the blue HandiHaler® and one actuation from the placebo MDPI in the morning and one actuation from the placebo MDPI in the evening.
  Period 2:
  18 µg Tiotropium (T18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® in the morning plus one actuation of 50 µg Salmeterol MDPI (S_DPI) BID, in the morning and in the evening, and one placebo capsule from blue Handi Haler® in the morning.
  Period 3: Fixed-dose combination of 7.5 µg/ 25 µg Tiotropium/Salmeterol (T+S_PE) inhalation powder from one capsule via the blue HandiHaler® once daily (QD) in the morning, one capsule of matching placebo via the grey HandiHaler® and one actuation from the placebo Multi-Dose Powder Inhaler (MDPI) in the morning and one actuation from the placebo MDPI in the evening.
  Period 4: One actuation of 50 µg Salmeterol MDPI (Salm50DPI) twice daily (BID), in the morning and in the evening, one capsule of matching placebo from grey HandiHaler® and one capsule of matching placebo from the blue HandiHaler® in the morning. Each dose of study medication had to be taken approximately at the same time, with 12 hours between the evening and morning dose. Each treatment period was 6 weeks on average with no wash-out between the treatment periods.
- Salm50DPI/ T+S_PE/ T18GEL+S_DPI/ Tio18GEL: Period 1: One actuation of 50 µg Salmeterol MDPI (Salm50DPI) twice daily (BID), in the morning and in the evening, one capsule of matching placebo from grey HandiHaler® and one capsule of matching placebo from the blue HandiHaler® in the morning.
  Period 2: Fixed-dose combination of 7.5 µg/ 25 µg Tiotropium/Salmeterol (T+S_PE) inhalation powder from one capsule via the blue HandiHaler® once daily (QD) in the morning, one capsule of matching placebo via the grey HandiHaler® and one actuation from the placebo Multi-Dose Powder Inhaler (MDPI) in the morning and one actuation from the placebo MDPI in the evening.
  Period 3: 18 µg Tiotropium (T18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® in the morning plus one actuation of 50 µg Salmeterol MDPI (S_DPI) BID, in the morning and in the evening, and one placebo capsule from blue Handi Haler® in the morning.
  Period 4: 18 µg Tiotropium (Tio18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® QD in the morning, one capsule of matching placebo via the blue HandiHaler® and one actuation from the placebo MDPI in the morning and one actuation from the placebo MDPI in the evening. Each dose of study medication had to be taken approximately at the same time, with 12 hours between the evening and morning dose. Each treatment period was 6 weeks on average with no wash-out between the treatment periods.
- T18GEL+S_DPI/ Salm50DPI/ Tio18GEL/ T+S_PE: Period 1: 18 µg Tiotropium (T18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® in the morning plus one actuation of 50 µg Salmeterol MDPI (S_DPI) BID, in the morning and in the evening, and one placebo capsule from blue Handi Haler® in the morning. Period 2: One actuation of 50 µg Salmeterol MDPI (Salm50DPI) twice daily (BID), in the morning and in the evening, one capsule of matching placebo from grey HandiHaler® and one capsule of matching placebo from the blue HandiHaler® in the morning. Period 3: 18 µg Tiotropium (Tio18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® QD in the morning, one capsule of matching placebo via the blue HandiHaler® and one actuation from the placebo MDPI in the morning and one actuation from the placebo MDPI in the evening. Period 4: Fixed-dose combination of 7.5 µg/ 25 µg Tiotropium/Salmeterol (T+S_PE) inhalation powder from one capsule via the blue HandiHaler® once daily (QD) in the morning, one capsule of matching placebo via the grey HandiHaler® and one actuation from the placebo Multi-Dose Powder Inhaler (MDPI) in the morning and one actuation from the placebo MDPI in the evening. Each dose of study medication had to be taken approximately at the same time, with 12 hours between the evening and morning dose. Each treatment period was 6 weeks on average with no wash-out between the treatment periods.
Period: Period 1
Arm/Group | T+S_PE/ Tio18GEL / Salm50DPI / T18GEL+S_DPI | Tio18GEL/ T18GEL+S_DPI/ T+S_PE/ Salm50DPI | Salm50DPI/ T+S_PE/ T18GEL+S_DPI/ Tio18GEL | T18GEL+S_DPI/ Salm50DPI/ Tio18GEL/ T+S_PE
Started | 34 | 38 | 36 | 39
Treated | 34 | 37 | 36 | 39
Completed (Not prematurely discontinued study medication) | 32 | 31 | 32 | 39
Not Completed | 2 | 7 | 4 | 0
Not completed — Personal Reasons | 0 | 0 | 1 | 0
Not completed — Refused continuing medication | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Other adverse event (AE) | 0 | 2 | 0 | 0
Not completed — Worsening of disease under study (AE) | 1 | 3 | 2 | 0
Not completed — Not treated | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | T+S_PE/ Tio18GEL / Salm50DPI / T18GEL+S_DPI | Tio18GEL/ T18GEL+S_DPI/ T+S_PE/ Salm50DPI | Salm50DPI/ T+S_PE/ T18GEL+S_DPI/ Tio18GEL | T18GEL+S_DPI/ Salm50DPI/ Tio18GEL/ T+S_PE
Started | 32 | 31 | 32 | 39
Treated | 32 | 31 | 32 | 39
Completed (Not prematurely discontinued from study medication) | 31 | 31 | 32 | 36
Not Completed | 1 | 0 | 0 | 3
Not completed — Worsening of disease under study | 1 | 0 | 0 | 3
Period: Period 3
Arm/Group | T+S_PE/ Tio18GEL / Salm50DPI / T18GEL+S_DPI | Tio18GEL/ T18GEL+S_DPI/ T+S_PE/ Salm50DPI | Salm50DPI/ T+S_PE/ T18GEL+S_DPI/ Tio18GEL | T18GEL+S_DPI/ Salm50DPI/ Tio18GEL/ T+S_PE
Started | 31 | 31 | 32 | 36
Treated | 31 | 31 | 32 | 36
Completed (Not prematurely discontinued from study medication) | 30 | 31 | 30 | 35
Not Completed | 1 | 0 | 2 | 1
Not completed — Refused continuing medication | 1 | 0 | 1 | 0
Not completed — Other adverse event (AE) | 0 | 0 | 1 | 1
Period: Period 4
Arm/Group | T+S_PE/ Tio18GEL / Salm50DPI / T18GEL+S_DPI | Tio18GEL/ T18GEL+S_DPI/ T+S_PE/ Salm50DPI | Salm50DPI/ T+S_PE/ T18GEL+S_DPI/ Tio18GEL | T18GEL+S_DPI/ Salm50DPI/ Tio18GEL/ T+S_PE
Started | 30 | 31 | 30 | 35
Treated | 30 | 31 | 30 | 35
Completed (Not prematurely discontinued from study medication) | 29 | 30 | 30 | 34
Not Completed | 1 | 1 | 0 | 1
Not completed — Refused continuing medication | 0 | 1 | 0 | 0
Not completed — Other adverse event (AE) | 1 | 0 | 0 | 0
Not completed — Worsening of disease under study (AE) | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set: All randomised patients who took at least one dose of study medication.
Groups:
- Study Total: Total number of patients treated in the study. This was a randomized, double-blind 4-way cross over study. Patients were assigned randomly to one of 4 treatment sequences in which they received each of the 4 treatments (7.5 µg/25 µg Tio/Salmeterol, 18 µg Tiotropium, 50 µg Salmeterol MDPI and 18 µg Tiotropium Free combination). The duration of each treatment period was 6 weeks on average with no washout period between treatments.
Arm/Group | Study Total
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 143
  More than one race | 0
  Unknown or Not Reported | 0
FEV1 AUC0-12 at baseline [Mean (Standard Deviation); unit: Liter (L)] — FEV1 AUC was defined as the area under the FEV1 curve normalized for time. It was calculated from time 0 to 12 h (FEV1 AUC0-12), using the trapezoidal rule divided by the corresponding duration (12 h) to give the results in liter (L). FEV1 AUC0-12 at baseline is reported. Population: Full Analysis Set (FAS): All patients where baseline data and any on-treatment efficacy data are available.
  Liter (L)
    number analyzed (Participants) | 135
    (all) | 1.55 (0.51)

OUTCOME MEASURES:

1. Primary Outcome: Response in Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve From 0 - 12 Hours (AUC0-12)
Description: FEV1 AUC was defined as the area under the FEV1 curve normalized for time. It was calculated from time 0 to 12 h (FEV1 AUC0-12), using the trapezoidal rule divided by the corresponding duration (12 h) to give the results in liter (L). FEV1 AUC0-12h response is defined as the change from baseline:
  FEV1 AUC0-12h response = FEV1 AUC0-12h - FEV1 (Baseline). The FEV1 baseline value is defined as the pre-dose FEV1 measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and 10 minutes (min) prior to inhalation and 30 min, 60 min, 2, 3, 4, 6, 8, 10 and 12 hours after inhalation of the morning dose after 6 weeks of treatment.
Population: Full Analysis Set (FAS): All patients where baseline data and any on-treatment efficacy data are available. This definition was applied separately for each endpoint, so that the number of patients analysed may vary across endpoints.
Measure: Mean (Standard Error); unit: Liter (L)
Groups:
- 7.5 µg /25 µg Tio /Salmeterol (T+S_PE): Fixed-dose combination of 7.5 µg/ 25 µg Tiotropium/Salmeterol (T+S_PE) inhalation powder from one capsule via the blue HandiHaler® once daily (QD) in the morning, one capsule of matching placebo via the grey HandiHaler® and one actuation from the placebo Multi-Dose Powder Inhaler (MDPI) in the morning and one actuation from the placebo MDPI in the evening. Each dose of study medication had to be taken approximately at the same time, with 12 hours between the evening and morning dose. Each treatment period was 6 weeks on average with no wash-out between the treatment periods.
- 18 µg Tiotropium (Tio18GEL): 18 µg Tiotropium (Tio18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® QD in the morning, one capsule of matching placebo via the blue HandiHaler® and one actuation from the placebo MDPI in the morning and one actuation from the placebo MDPI in the evening. Each dose of study medication had to be taken approximately at the same time, with 12 hours between the evening and morning dose. Each treatment period was 6 weeks on average with no wash-out between the treatment periods.
- 50 µg Salmeterol MDPI (Salm50DPI): One actuation of 50 µg Salmeterol MDPI (Salm50DPI) twice daily (BID) in the morning and in the evening, one capsule of matching placebo from grey HandiHaler® and one capsule of matching placebo from the blue HandiHaler® in the morning. Each dose of study medication had to be taken approximately at the same time, with 12 hours between the evening and morning dose. Each treatment period was 6 weeks on average with no wash-out between the treatment periods.
- 18 µg Tiotropium Free Combination (T18GEL+S_DPI): 18 µg Tiotropium (T18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® in the morning plus one actuation of 50 µg Salmeterol MDPI (S_DPI) BID, in the morning and in the evening, and one placebo capsule from blue Handi Haler® in the morning. Each dose of study medication had to be taken approximately at the same time, with 12 hours between the evening and morning dose. Each treatment period was 6 weeks on average with no wash-out between the treatment periods.
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter (L) | 0.187 (0.026) | 0.117 (0.026) | 0.057 (0.026) | 0.211 (0.026)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); H1: Superiority of FDC Tiotropium/Salmeterol (T+S_PE) vs. salmeterol (Salm50DPI) for FEV1 AUC0-12; Test type: Superiority; p < 0.0001, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period; Difference of adjusted means = 0.130, 95% CI 2-sided [0.102 to 0.158], Standard Error of Mean 0.014 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); H1: Superiority of FDC Tiotropium/Salmeterol (T+S_PE) vs Tiotropium (Tio18GEL) for FEV1 AUC0- 12; Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Difference of adjusted means = 0.070, 95% CI 2-sided [0.042 to 0.097], Standard Error of Mean 0.014 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); The Tiotropium free combination (T18GEL+S_DPI) was included in order to characterise this treatment in comparison with the FDC Tiotropium/Salmeterol (T+S_PE). No formal hypotheses were defined; Test type: Other; p = 0.0914, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Difference of adjusted means = -0.024, 95% CI 2-sided [-0.052 to 0.004], Standard Error of Mean 0.014 — (T+S_PE) - (T18GEL+S-DPI)

2. Primary Outcome: Response in Forced Expiratory Volume in Second (FEV1) Area Under the Curve From 12 - 24 Hours (AUC12 -24)
Description: The FEV1 AUC was defined as the area under the FEV1 curve (AUC) normalised for time. It was calculated from time 12 to 24 h (FEV1 AUC12-24), using the trapezoidal rule divided by the corresponding duration (i.e. 12 h) to give the results in L.
  AUC12-24h response is defined as the change from baseline:
  FEV1 AUC12-24h response = FEV1 AUC12-24h - FEV1 (Baseline). The FEV1 baseline value is defined as the pre-dose FEV1 measurement in the morning at the randomization visit (Visit 2) just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and 10 minutes (min) prior to inhalation and 30 min, 60 min, 2, 10, 11, and 12 hours after inhalation of the evening dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter (L)
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter (L) | 0.068 (0.025) | 0.003 (0.025) | 0.003 (0.025) | 0.124 (0.025)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); H1: Non-Inferiority of FDC Tiotropium/Salmeterol (T+S_PE) vs. Salmeterol (Salm50DPI) for FEV1AUC12-24; Test type: Non-Inferiority — The non-inferiority margin for FEV1 endpoints was defined as d=0.050 L; p < .0001, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Difference of adjusted means = 0.064, 95% CI 2-sided [0.036 to 0.093], Standard Error of Mean 0.015 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); H1: Non-inferiority of FDC Tiotropium/Salmeterol (T+S_PE) vs. Tiotropium (TIO18GEL) of FEV1AUC12-24; Test type: Non-Inferiority — The non-inferiority margin for FEV1 endpoints was defined as d=0.050 L; p < .0001, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Difference of adjusted means = 0.064, 95% CI 2-sided [0.036 to 0.093], Standard Error of Mean 0.015 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.0001, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Difference of adjusted means = -0.057, 95% CI 2-sided [-0.086 to -0.028], Standard Error of Mean 0.015 — (T+S_PE) - (T18GEL+S-DPI)

3. Primary Outcome: Response in Peak Forced Expiratory Volume in 1 Second (FEV1)
Description: Peak FEV1 was defined as the highest FEV1 reading observed within 3 hours after inhalation of the last morning dose of each randomized treatment. Peak FEV1 response is defined as change from baseline:
  Peak FEV1 response = Peak FEV1 - FEV1 (Baseline). The FEV1 baseline value is defined as the pre-dose FEV1 measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and within 3 hours post-morning dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter
Groups:
- 18µg Tiotropium (Tio18GEL): 18 µg Tiotropium (Tio18GEL) inhalation powder from one capsule via the grey Spiriva HandyHaler® QD in the morning, one capsule of matching placebo via the blue HandiHaler® and one actuation from the placebo MDPI in the morning and one actuation from the placebo MDPI in the evening. Each dose of study medication had to be taken approximately at the same time, with 12 hours between the evening and morning dose. Each treatment period was 6 weeks on average with no wash-out between the treatment periods.
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter | 0.296 (0.026) | 0.229 (0.026) | 0.161 (0.026) | 0.320 (0.026)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); H1: Superiority of FDC Tiotropium/Salmeterol (T+S_PE) vs. Salmeterol (Salm50DPI) of Peak FEV1; Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Difference of adjusted means = 0.134, 95% CI 2-sided [0.102 to 0.166], Standard Error of Mean 0.016 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); H1: Superiority of FDC Tiotropium/Salmeterol (T+S_PE) vs. Tiotropium (TIO18GEL) of PeakFEV1; Test type: Superiority; p < .0001, ANOVA; Analysis of with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Difference of adjusted means = 0.066, 95% CI 2-sided [0.034 to 0.098], Standard Error of Mean 0.016 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.1093, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Difference of adjusted means = -0.026, 95% CI 2-sided [-0.058 to 0.006], Standard Error of Mean 0.016 — (T+S_PE) - (T18GEL+S_DPI)

4. Primary Outcome: Response in Trough Forced Expiratory Volume in 1 Second (FEV1)
Description: Trough FEV1 is determined at the end of each treatment period and is defined as the pre-dose FEV1 measured just prior to the last administration of the morning dose of randomized treatment.
  Trough FEV1 response is defined as the change from baseline:
  Trough FEV1 response = Trough FEV1 - FEV1 (Baseline) The FEV1 baseline value is defined as the pre-dose FEV1 measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and 5 minutes prior to the last administration of the morning dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter | 0.062 (0.024) | 0.032 (0.024) | 0.003 (0.024) | 0.097 (0.024)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); H1: Non-inferiority of FDC Tiotropium/Salmeterol (T+S_PE) vs. Salmeterol (Salm50DPI) of trough FEV1; Test type: Non-Inferiority — The non-inferiority margin for FEV1 endpoints was defined as d=0.050 L; p = 0.0008, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Differences of adjusted means = 0.058, 95% CI 2-sided [0.024 to 0.092], Standard Error of Mean 0.017 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); H1: Non-inferiority of FDC Tiotropium/Salmeterol (T+S_PE) vs. Tiotropium (TIO18GEL) of trough FEV1; Test type: Non-Inferiority — The non-inferiority margin for FEV1 endpoints was defined as a delta of 0.050 L; p = 0.0857, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Difference of adjusted means = 0.029, 95% CI 2-sided [-0.004 to 0.063], Standard Error of Mean 0.017 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.0317, ANOVA; Analysis of variance with terms for centre, patient with centre, treatment, and period. α = 0.025 one-sided; Difference of adjusted means = -0.037, 95% CI 2-sided [-0.071 to -0.003], Standard Error of Mean 0.017 — (T+S_PE) - (T18GEL+S-DPI)

5. Secondary Outcome: Response in Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve From 0-24 Hours (AUC0-24)
Description: FEV1 AUC was defined as the area under the FEV1 curve normalized for time. It was calculated from time 0 to 24 h (FEV1 AUC0-24), using the trapezoidal rule divided by the corresponding duration (24 h) to give the results in liter (L). FEV1 AUC0-24h response is defined as the change from baseline:
  FEV1 AUC0-24h response = FEV1 AUC0-24h - FEV1 (Baseline). The FEV1 baseline value is defined as the pre-dose FEV1 measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and 10 minutes (min) prior and 60 min, 2, 3, 4, 6, 8, 10 and 12 hours after inhalation of the morning dose and 30 min, 60 min, 2, 10, 11, and 12 hours after inhalation of the evening dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter | 0.128 (0.025) | 0.060 (0.025) | 0.030 (0.025) | 0.167 (0.025)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); H1: Superiority of FDC Tiotropium/Salmeterol (T+S_PE) vs. salmeterol (Salm50DPI) for FEV1 AUC0-24; Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.097, 95% CI 2-sided [0.071 to 0.124], Standard Error of Mean 0.014 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); H1: Superiority of FDC Tiotropium/Salmeterol (T+S_PE) vs. Tiotropium (TIO18GEL) for FEV1 AUC24; Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted mean difference = 0.067, 95% CI 2-sided [0.041 to 0.093], Standard Error of Mean 0.013 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.0029, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.041, 95% CI 2-sided [-0.067 to -0.014], Standard Error of Mean 0.014 — (T+S_PE) - (T18GEL+S-DPI)

6. Secondary Outcome: Response in Forced Vital Capacity (FVC) Area Under the Curve From 0 to 12 Hours (AUC0-12)
Description: FVC AUC was defined as the area under the FVC curve normalized for time. It was calculated from time 0 to 12 h (FVC AUC0-12), using the trapezoidal rule divided by the corresponding duration (12 h) to give the results in liter (L). FVC AUC0-12h response is defined as the change from baseline:
  FVC AUC0-12h response = FVC AUC0-12h - FVC (Baseline). The baseline value for FVC based parameters is defined as the pre-dose FVC measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter | 0.337 (0.047) | 0.253 (0.047) | 0.160 (0.048) | 0.381 (0.047)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.0010, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.083, 95% CI 2-sided [0.034 to 0.132], Standard Error of Mean 0.025 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.176, 95% CI 2-sided [0.127 to 0.226], Standard Error of Mean 0.025 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.0757, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.045, 95% CI 2-sided [-0.095 to 0.005], Standard Error of Mean 0.025 — (T+S_PE) - (T18GEL+S-DPI)

7. Secondary Outcome: Response in Forced Vital Capacity (FVC) Area Under the Curve From 12 to 24 Hours (AUC12-24)
Description: The FVC AUC was defined as the area under the FVC curve (AUC) normalised for time. It was calculated from time 12 to 24 h (FVC AUC12-24), using the trapezoidal rule divided by the corresponding duration (i.e. 12 h) to give the results in L.
  AUC12-24h response is defined as the change from baseline:
  FVC AUC12-24h response = FVC AUC12-24h - FVC (Baseline). The FVC baseline value is defined as the pre-dose FVC measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and 10 minutes (min) prior to inhalation and 30 min, 60 min, 2, 10, 11 and 12 hours after inhalation of the evening dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter | 0.163 (0.048) | 0.076 (0.048) | 0.043 (0.048) | 0.245 (0.048)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.0015, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.085, 95% CI 2-sided [0.033 to 0.137], Standard Error of Mean 0.027 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.118, 95% CI 2-sided [0.066 to 0.171], Standard Error of Mean 0.027 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.0017, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.085, 95% CI 2-sided [-0.138 to -0.032], Standard Error of Mean 0.027 — (T+S_PE) - (T18GEL+S-DPI)

8. Secondary Outcome: Response in Forced Vital Capacity (FVC) Area Under the Curve From 0 - 24 Hours (AUC0-24)
Description: The FVC AUC was defined as the area under the FVC curve (AUC) normalised for time. It was calculated from time 0 to 24 h (FVC AUC0-24), using the trapezoidal rule divided by the corresponding duration (i.e. 24 h) to give the results in L. AUC response was defined as the change from the baseline FVC; baseline was defined as the FVC measured on randomisation visit. Mean is adjusted mean.
Time Frame: At baseline and 10 minutes (min) prior and 60 min, 2, 3, 4, 6, 8, 10 and 12 hour after inhalation the morning dose and 30 min, 60 min, 2, 10, 11, and 12 hours after inhalation of the evening dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter | 0.250 (0.046) | 0.165 (0.046) | 0.102 (0.046) | 0.313 (0.046)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.0005, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.084, 95% CI 2-sided [0.037 to 0.131], Standard Error of Mean 0.024 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.147, 95% CI 2-sided [0.100 to 0.194], Standard Error of Mean 0.024 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.0074, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.065, 95% CI 2-sided [-0.113 to -0.018], Standard Error of Mean 0.024 — (T+S_PE) - (T18GEL+S-DPI)

9. Secondary Outcome: Response in Peak Forced Vital Capacity (FVC)
Description: as for outcome 3
Time Frame: At baseline and within 3 hours post-morning dose after 6 weeks of treatment.
Population: Full Analysis Set (FAS): All patients where baseline data and any on-treatment efficacy data are available. This definition was applied separately for each endpoint, so that the number of patients analyzed may vary across endpoints.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter | 0.502 (0.049) | 0.449 (0.049) | 0.359 (0.050) | 0.556 (0.049)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.0898, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Differences of adjusted means = 0.051, 95% CI 2-sided [-0.008 to 0.109], Standard Error of Mean 0.030 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.142, 95% CI 2-sided [0.083 to 0.201], Standard Error of Mean 0.030 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.0601, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.057, 95% CI 2-sided [-0.116 to 0.002], Standard Error of Mean 0.030 — (T+S_PE) - (T18GEL+S-DPI)

10. Secondary Outcome: Response in Trough Forced Vital Capacity (FVC)
Description: Trough FVC1 is determined at the end of each 6-week treatment period and is defined as the pre-dose FVC1 measured just prior to the last administration of the morning dose of randomized treatment.
  Trough FVC1 response is defined as the change from baseline:
  Trough FVC1 response = Trough FVC1 - FVC1 (Baseline) The FVC1 baseline value is defined as the pre-dose FVC1 measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and 5 minutes prior to the last administration of the morning dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter | 0.139 (0.047) | 0.165 (0.047) | 0.095 (0.048) | 0.229 (0.047)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.3652, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.028, 95% CI 2-sided [-0.089 to 0.033], Standard Error of Mean 0.031 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p = 0.1816, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.042, 95% CI 2-sided [-0.020 to 0.103], Standard Error of Mean 0.031 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.0026, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.095, 95% CI 2-sided [-0.157 to -0.033], Standard Error of Mean 0.031 — (T+S_PE) - (T18GEL+S-DPI)

11. Secondary Outcome: Response in Peak Expiratory Flow Rate (PEF) Area Under the Curve Form 0 to 12 Hours (AUC0-12)
Description: PEF(L/min) AUC0-12(h) response is defined as the change from baseline. AUC0-12(h) was calculated as the area under the curve from 0 to 12 hours using the trapezoidal rule, divided by the full duration (12 hours) to report in liter/minutes.
  PEF AUC0-12h response = PEF AUC0-12h - PEF (Baseline). The PEF baseline value is defined as the pre-dose PEF measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and 10 minutes (min) prior and 30 min, 60 min, 2, 3, 4, 6, 8, 10 and 12 hours after inhalation of the morning dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter/minutes (L/min)
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter/minutes (L/min) | 34.5 (5.2) | 22.5 (5.2) | 10.2 (5.2) | 37.8 (5.1)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 11.8, 95% CI 2-sided [6.9 to 16.8], Standard Error of Mean 2.5 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 24.2, 95% CI 2-sided [19.2 to 29.2], Standard Error of Mean 2.5 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.1804, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -3.4, 95% CI 2-sided [-8.5 to 1.6], Standard Error of Mean 2.6 — (T+S_PE) - (T18GEL+S-DPI)

12. Secondary Outcome: Response in Peak Expiratory Flow Rate (PEF) Area Under the Curve From 12 to 24 Hours (AUC12-24)
Description: PEF(L/min) AUC12-24(h) response is defined as the change from baseline. AUC12-24(h) was calculated as the area under the curve from 12 to 24 hours using the trapezoidal rule, divided by the full duration (12 hours) to report in liter/minutes.
  PEF AUC12-24h response = PEF AUC12-24h - PEF (Baseline). The PEF baseline value is defined as the pre-dose PEF measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and 10 minutes (min) prior and 30 min, 60 min, 2, 10, 11 and 12 hours after inhalation of the evening dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter/minutes (L/min)
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter/minutes (L/min) | 7.3 (5.1) | -1.3 (5.1) | -3.4 (5.1) | 20.0 (5.1)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.0008, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 8.5, 95% CI 2-sided [3.5 to 13.4], Standard Error of Mean 2.5 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 10.6, 95% CI 2-sided [5.6 to 15.5], Standard Error of Mean 2.5 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -12.9, 95% CI 2-sided [-17.9 to -8.0], Standard Error of Mean 2.5 — (T+S_PE) - (T18GEL+S_DPI)

13. Secondary Outcome: Response in Peak Expiratory Flow Rate (PEF) Area Under the Curve From 0 to 24 Hours (AUC0-24)
Description: PEF(L/min) AUC0-24(h) response is defined as the change from baseline. AUC0-24(h) was calculated as the area under the curve from 0 to 24 hours using the trapezoidal rule, divided by the full duration (24 hours) to report in liter/minutes.
  PEF AUC0-24h response = PEF AUC0-24h - PEF (Baseline). The PEF baseline value is defined as the pre-dose PEF measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter/minutes (L/min)
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter/minutes (L/min) | 20.8 (5.0) | 10.6 (5.0) | 3.4 (5.0) | 28.9 (5.0)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 10.1, 95% CI 2-sided [5.7 to 14.6], Standard Error of Mean 2.3 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 17.4, 95% CI 2-sided [12.9 to 21.9], Standard Error of Mean 2.3 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.0004, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -8.2, 95% CI 2-sided [-12.7 to -3.7], Standard Error of Mean 2.3 — (T+S_PE) - (T18GEL+S_DPI)

14. Secondary Outcome: Response in Peak PEF (Peak Expiratory Flow Rate)
Description: Peak PEF was defined as the highest PEF reading observed within 3 hours after inhalation of the last morning dose of randomized treatment.
  Peak PEF response is defined as change from baseline:
  Peak PEF response = Peak PEF - PEF (Baseline). The PEF baseline value is defined as the pre-dose PEF measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and within 3 hours post-morning dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter/minutes (L/min)
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter/minutes (L/min) | 53.9 (5.2) | 40.6 (5.2) | 30.8 (5.3) | 59.0 (5.2)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 13.1, 95% CI 2-sided [7.2 to 18.9], Standard Error of Mean 3.0 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 23.1, 95% CI 2-sided [17.2 to 28.9], Standard Error of Mean 3.0 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.0769, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference in adjusted means = -5.3, 95% CI 2-sided [-11.2 to 0.6], Standard Error of Mean 3.0 — (T+S_PE) - (T18GEL+S-DPI)

15. Secondary Outcome: Response in Trough Peak Expiratory Flow Rate (PEF)
Description: Trough PEF is determined at the end of each treatment period and is defined as the pre-dose PEF measured just prior to the last administration of the morning dose of randomized treatment. Trough PEF response is defined as the change from baseline:
  Trough PEF response = Trough PEF - PEF (Baseline) The PEF baseline value is defined as the pre-dose PEF measurement in the morning at the randomization visit just prior to administration of the first dose of randomized treatment. Mean is adjusted mean.
Time Frame: At baseline and 5 minutes prior to the last administration of the morning dose after 6 weeks of treatment.
Population: Full Analysis Set: All patients where baseline data and any on-treatment efficacy data are available. This definition was applied separately for each endpoint, so that the number of patients analysed may vary across endpoints.
Measure: Mean (Standard Error); unit: Liter/minutes (L/min)
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter/minutes (L/min) | 14.4 (4.9) | 11.3 (4.9) | 7.1 (4.9) | 22.9 (4.9)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.3775, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 2.8, 95% CI 2-sided [-3.5 to 9.1], Standard Error of Mean 3.2 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p = 0.0285, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 7.1, 95% CI 2-sided [0.7 to 13.4], Standard Error of Mean 3.2 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.0065, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -8.9, 95% CI 2-sided [-15.2 to -2.5], Standard Error of Mean 3.2 — (T+S_PE) - (T18GEL+S-DPI)

16. Secondary Outcome: Response in Individual Forced Expiratory Volume in 1 Second (FEV1) Over a 24 Hour Observation Period
Description: Response in individual forced expiratory volume in 1 second (FEV1) over a 24 hour observation period. Response is defined as change from baseline.
  Means are adjusted for treatment, centre, treatment period and patient within centre.
Time Frame: At baseline, pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 12.5, 13, 14, 22, 23, and 24 hours post morning dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter (L)
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter (L)
  0 hour | 0.062 (0.024) | 0.032 (0.024) | 0.003 (0.024) | 0.097 (0.024)
  0.5 hour | 0.180 (0.024) | 0.129 (0.024) | 0.068 (0.025) | 0.204 (0.024)
  1 hour | 0.211 (0.025) | 0.139 (0.025) | 0.084 (0.025) | 0.236 (0.025)
  2 hour | 0.242 (0.026) | 0.163 (0.026) | 0.108 (0.026) | 0.277 (0.026)
  3 hour | 0.257 (0.027) | 0.167 (0.027) | 0.111 (0.027) | 0.277 (0.027)
  4 hour | 0.231 (0.027) | 0.162 (0.027) | 0.102 (0.027) | 0.262 (0.027)
  6 hour | 0.209 (0.028) | 0.121 (0.028) | 0.064 (0.028) | 0.218 (0.028)
  8 hour | 0.167 (0.028) | 0.098 (0.028) | 0.044 (0.028) | 0.185 (0.028)
  10 hour | 0.138 (0.028) | 0.080 (0.028) | 0.006 (0.028) | 0.166 (0.028)
  12 hour | 0.117 (0.027) | 0.060 (0.027) | -0.007 (0.027) | 0.137 (0.027)
  12.5 hour | 0.101 (0.028) | 0.048 (0.028) | 0.021 (0.028) | 0.147 (0.028)
  13 hour | 0.105 (0.028) | 0.043 (0.028) | 0.035 (0.028) | 0.153 (0.028)
  14 hour | 0.115 (0.029) | 0.040 (0.029) | 0.031 (0.029) | 0.172 (0.028)
  22 hour | 0.005 (0.025) | -0.057 (0.025) | -0.034 (0.025) | 0.068 (0.025)
  23 hour | 0.071 (0.025) | 0.018 (0.025) | 0.008 (0.026) | 0.116 (0.025)
  24 hour | 0.112 (0.025) | 0.058 (0.025) | 0.024 (0.026) | 0.147 (0.025)

17. Secondary Outcome: Response in Individual Forced Vital Capacity (FVC) Over a 24 Hour Observation Period
Description: Response in forced vital capacity (FVC) over a 24 hour observation period. Response is defined as change from baseline.
Time Frame: At baseline, pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 12.5, 13, 14, 22, 23 and 24 hours post morning dose after 6 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter
  0 hour | 0.139 (0.047) | 0.165 (0.047) | 0.095 (0.048) | 0.229 (0.047)
  0.5 hour | 0.354 (0.049) | 0.302 (0.049) | 0.200 (0.049) | 0.395 (0.048)
  1 hour | 0.386 (0.050) | 0.332 (0.050) | 0.220 (0.050) | 0.411 (0.050)
  2 hours | 0.409 (0.049) | 0.330 (0.049) | 0.243 (0.050) | 0.464 (0.049)
  3 hours | 0.425 (0.051) | 0.319 (0.051) | 0.252 (0.051) | 0.457 (0.051)
  4 hours | 0.396 (0.050) | 0.312 (0.050) | 0.223 (0.050) | 0.463 (0.050)
  6 hours | 0.368 (0.050) | 0.254 (0.051) | 0.179 (0.051) | 0.399 (0.050)
  8 hours | 0.309 (0.051) | 0.225 (0.051) | 0.141 (0.051) | 0.355 (0.051)
  10 hours | 0.264 (0.051) | 0.185 (0.051) | 0.051 (0.051) | 0.306 (0.051)
  12 hours | 0.229 (0.050) | 0.142 (0.050) | 0.051 (0.051) | 0.258 (0.050)
  12.5 hours | 0.206 (0.052) | 0.131 (0.053) | 0.066 (0.053) | 0.273 (0.052)
  13 hours | 0.194 (0.052) | 0.116 (0.052) | 0.106 (0.052) | 0.266 (0.052)
  14 hours | 0.225 (0.052) | 0.122 (0.052) | 0.082 (0.052) | 0.287 (0.052)
  22 hours | 0.081 (0.049) | 0.001 (0.049) | -0.014 (0.049) | 0.191 (0.049)
  23 hours | 0.176 (0.050) | 0.098 (0.050) | 0.043 (0.050) | 0.243 (0.050)
  24 hours | 0.208 (0.050) | 0.153 (0.050) | 0.089 (0.050) | 0.280 (0.050)

18. Secondary Outcome: Response in Individual Peak Expiratory Flow (PEF) Over a 24 Hour Observation Period
Description: Response in individual peak expiratory flow (PEF) over a 24 hour observation period. Response is defined as change from baseline.
  Means are adjusted for treatment, centre, treatment period and patient within centre.
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter/minutes (L/min)
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Liter/minutes (L/min)
  0 hour | 14.4 (4.9) | 11.3 (4.9) | 7.1 (4.9) | 22.9 (4.9)
  0.5 hour | 30.8 (5.1) | 20.1 (5.2) | 13.7 (5.2) | 34.3 (5.1)
  1 hour | 35.5 (5.1) | 22.2 (5.1) | 14.6 (5.1) | 41.0 (5.1)
  2 hours | 42.2 (5.3) | 27.6 (5.3) | 18.5 (5.3) | 47.0 (5.2)
  3 hours | 45.0 (5.4) | 27.9 (5.4) | 17.1 (5.4) | 49.9 (5.4)
  4 hours | 41.9 (5.6) | 26.4 (5.6) | 17.2 (5.6) | 46.5 (5.5)
  6 hours | 37.8 (5.5) | 25.0 (5.5) | 11.1 (5.5) | 38.9 (5.5)
  8 hours | 33.9 (5.6) | 23.3 (5.6) | 8.6 (5.6) | 35.5 (5.6)
  10 hours | 26.9 (5.7) | 19.0 (5.7) | 1.9 (5.7) | 28.8 (5.7)
  12 hours | 23.4 (5.6) | 11.8 (5.6) | -0.6 (5.6) | 26.8 (5.6)
  12.5 hours | 13.6 (5.7) | 5.5 (5.7) | -0.7 (5.8) | 26.6 (5.7)
  13 hours | 12.0 (5.7) | 5.8 (5.7) | 2.6 (5.7) | 25.3 (5.6)
  14 hours | 15.6 (5.7) | 4.5 (5.7) | 1.4 (5.8) | 27.9 (5.7)
  22 hours | -4.2 (5.1) | -11.7 (5.1) | -9.7 (5.1) | 10.1 (5.1)
  23 hours | 9.1 (5.3) | 2.3 (5.3) | -5.7 (5.3) | 18.1 (5.3)
  24 hours | 14.0 (5.3) | 9.6 (5.3) | 2.0 (5.3) | 24.0 (5.3)

19. Secondary Outcome: Response in Morning and Evening Peak Expiratory Flow Rate (PEF), Recorded by Patients at Home
Description: The mean PEF is defined as the mean of the values obtained during the weeks after the first three weeks of treatment. Morning and evening mean PEF were calculated and analyzed separately. PEF was measured twice daily (in the morning prior to inhalation of study medication and in the evening prior to inhalation of study medication).
  Morning and evening mean PEF response are defined as the change from morning and evening baseline, respectively.
  Morning and evening mean PEF baseline are defined as the mean of the morning and evening values, respectively obtained from the last week preceding the randomization visit.
  Mean is adjusted for treatment, center, treatment period and patient within center.
Time Frame: At baseline and last 3 weeks of 6-week treatment period.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter / minute (L/min)
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 127 | 124 | 125
Liter / minute (L/min)
  PEF, morning | 6.8 (4.0) | 1.2 (4.0) | 0.6 (4.0) | 14.8 (4.0)
  PEF, evening: number analyzed (Participants) | 127 | 127 | 123 | 123
  PEF, evening | 16.7 (4.9) | 5.8 (4.9) | -6.4 (4.9) | 15.2 (4.9)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Morning PEF; Test type: Superiority; p = 0.0182, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 5.7, 95% CI 2-sided [1.0 to 10.4], Standard Error of Mean 2.4 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Morning PEF; Test type: Superiority; p = 0.0091, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 6.3, 95% CI 2-sided [1.6 to 11.1], Standard Error of Mean 2.4 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Morning PEF; Test type: Superiority; p = 0.0010, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -8.0, 95% CI 2-sided [-12.8 to -3.3], Standard Error of Mean 2.4 — (T+S_PE) - (T18GEL+S-DPI)
Statistical Analysis 4: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Evening PEF; Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 11.0, 95% CI 2-sided [5.8 to 16.2], Standard Error of Mean 2.6 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 5: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Evening PEF; Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 23.3, 95% CI 2-sided [18.1 to 28.6], Standard Error of Mean 2.7 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 6: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Evening PEF; Test type: Superiority; p = 0.5766, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 1.5, 95% CI 2-sided [-3.8 to 6.8], Standard Error of Mean 2.7 — (T+S_PE) - (T18GEL+S-DPI)

20. Secondary Outcome: Response in Morning and Evening Forced Expiratory Volume in 1 Second (FEV1) Recorded by Participants at Home
Description: Per treatment period, the morning mean FEV1 (mean of the pre-dose morning FEV1 measurements) and evening mean FEV1 (mean of the pre-dose evening FEV1 measurement) were calculated. Per treatment period the data obtained after the first 3 weeks were used for calculating these means.
  Morning and evening mean FEV1 responses are defined as the change from morning and evening baseline, respectively. The baseline values, morning and evening mean FEV1(Baseline), are defined as the mean of the morning and evening values, respectively obtained from the last week preceding the randomization visit .
  Mean is adjusted for treatment, centre, treatment period and patient within centre.
Time Frame: At baseline and last 3 weeks of 6-week treatment period.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Liter (L)
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 127 | 124 | 125
Liter (L)
  FEV1, morning | 0.052 (0.035) | 0.013 (0.035) | 0.026 (0.035) | 0.075 (0.035)
  FEV1, evening: number analyzed (Participants) | 127 | 127 | 123 | 123
  FEV1, evening | 0.094 (0.036) | 0.038 (0.036) | -0.010 (0.036) | 0.075 (0.036)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Morning FEV1; Test type: Superiority; p = 0.0137, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.040, 95% CI 2-sided [0.008 to 0.071], Standard Error of Mean 0.016 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Morning FEV1; Test type: Superiority; p = 0.0981, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.027, 95% CI 2-sided [-0.005 to 0.059], Standard Error of Mean 0.016 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Morning FEV1; Test type: Superiority; p = 0.1827, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.022, 95% CI 2-sided [-0.054 to 0.010], Standard Error of Mean 0.016 — (T+S_PE) - (T18GEL+S-DPI)
Statistical Analysis 4: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18µg Tiotropium (Tio18GEL); Evening FEV1; Test type: Superiority; p = 0.0014, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.057, 95% CI 2-sided [0.022 to 0.092], Standard Error of Mean 0.018 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 5: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Evening FEV1; Test type: Superiority; p < .0001, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.105, 95% CI 2-sided [0.070 to 0.140], Standard Error of Mean 0.018 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 6: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Evening FEV1; Test type: Superiority; p = 0.2584, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.020, 95% CI 2-sided [-0.015 to 0.056], Standard Error of Mean 0.018 — (T+S_PE) - (T18GEL+S-DPI)

21. Secondary Outcome: Response in Mean Number of Days With Rescue Medication Use
Description: Response (change from baseline) in mean number of days with rescue medication use in day-time, night-time and 24-hours. Per treatment period, the response in mean number of days using rescue medication was calculated for day-time (from inhalation of morning dose until 12 hours thereafter), night-time (from inhalation of evening dose until 12 hours thereafter) and 24h-total (from inhalation of morning dose until 24 hours thereafter) separately.
  Per 6-week treatment period the data obtained after the first 3 weeks was used for calculating means. Mean is adjusted mean.
Time Frame: At baseline and last 3 weeks of 6-week treatment period.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 127 | 124 | 125
Days
  Daytime | -0.08 (0.03) | -0.01 (0.03) | -0.06 (0.03) | -0.11 (0.03)
  Night-time: number analyzed (Participants) | 127 | 127 | 123 | 123
  Night-time | -0.15 (0.04) | -0.06 (0.04) | -0.07 (0.04) | -0.14 (0.04)
  24 hours: number analyzed (Participants) | 126 | 125 | 121 | 123
  24 hours | -0.13 (0.04) | -0.04 (0.04) | -0.06 (0.04) | -0.14 (0.04)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); Daytime; Test type: Superiority; p = 0.0027, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.07, 95% CI 2-sided [-0.11 to -0.02], Standard Error of Mean 0.02 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Daytime; Test type: Superiority; p = 0.4587, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.02, 95% CI 2-sided [-0.06 to 0.03], Standard Error of Mean 0.02 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Daytime; Test type: Superiority; p = 0.1535, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.03, 95% CI 2-sided [-0.01 to 0.08], Standard Error of Mean 0.02 — (T+S_PE) - (T18GEL+S-DPI)
Statistical Analysis 4: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); Night-time; Test type: Superiority; p = 0.0002, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.09, 95% CI 2-sided [-0.14 to -0.05], Standard Error of Mean 0.02 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 5: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Night-time; Test type: Superiority; p = 0.0006, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.09, 95% CI 2-sided [-0.14 to -0.04], Standard Error of Mean 0.03 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 6: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Night-time; Test type: Superiority; p = 0.5784, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.01, 95% CI 2-sided [-0.06 to 0.04], Standard Error of Mean 0.03 — (T+S_PE) - (T18GEL+S-DPI)
Statistical Analysis 7: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); 24 hours; Test type: Superiority; p = 0.0003, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.09, 95% CI 2-sided [-0.14 to -0.04], Standard Error of Mean 0.02 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 8: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); 24 hours; Test type: Superiority; p = 0.0042, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.07, 95% CI 2-sided [-0.12 to -0.02], Standard Error of Mean 0.02 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 9: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); 24 hours; Test type: Superiority; p = 0.9978, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.00, 95% CI 2-sided [-0.05 to 0.05], Standard Error of Mean 0.03 — (T+S_PE) - (T18GEL+S-DPI)

22. Secondary Outcome: Response in Mean Number of Puffs of Rescue Medication
Description: Response in mean number of puffs of rescue medication. Per treatment period, the response in mean number of puffs rescue medication used was calculated, for day-time (from inhalation of morning dose until 12 hours thereafter), night-time (from inhalation of evening dose until 12 hours thereafter) and 24h-total (from inhalation of morning dose until 24 hours thereafter) separately. Per 6-week treatment period the data obtained after the first 3 weeks was used for calculating means. Night-time, day-time and 24h-total mean number of puffs rescue medication used responses are defined as the change from night-time, day-time and 24h-total baseline, respectively.
  The baseline values, night-time, day-time and 24h-total mean mean number of puffs rescue medication used (Baseline), are defined as the mean of the night-time, day-time and 24h-total values, respectively obtained from the last week preceding the randomisation visit.
Time Frame: At baseline and last 3 weeks of 6-week treatment period.
Population: Full Analysis Set (FAS): All patients where baseline data any on-treatment efficacy data are available. This definition was applied separately for each endpoint, so that the number of patients analysed may vary across endpoints.
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Puffs
  Daytime: number analyzed (Participants) | 127 | 127 | 123 | 123
  Daytime | -0.61 (0.18) | -0.27 (0.18) | -0.25 (0.18) | -0.65 (0.18)
  Night-time: number analyzed (Participants) | 127 | 127 | 124 | 125
  Night-time | -0.16 (0.12) | 0.01 (0.12) | -0.07 (0.12) | -0.28 (0.12)
  Over 24 hours: number analyzed (Participants) | 126 | 125 | 121 | 123
  Over 24 hours | -0.76 (0.28) | -0.23 (0.28) | -0.30 (0.28) | -0.92 (0.28)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); Daytime; Test type: Superiority; p = 0.0029, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.33, 95% CI 2-sided [-0.55 to -0.11], Standard Error of Mean 0.11 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Daytime; Test type: Superiority; p = 0.0012, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.36, 95% CI 2-sided [-0.58 to -0.14], Standard Error of Mean 0.11 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Daytime; Test type: Superiority; p = 0.0829, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.12, 95% CI 2-sided [-0.02 to 0.25], Standard Error of Mean 0.07 — (T+S_PE) - (T18GEL+S-DPI)
Statistical Analysis 4: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); Night-time; Test type: Superiority; p = 0.0115, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.17, 95% CI 2-sided [-0.30 to -0.04], Standard Error of Mean 0.07 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 5: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Night-time; Test type: Superiority; p = 0.1772, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.09, 95% CI 2-sided [-0.22 to 0.04], Standard Error of Mean 0.07 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 6: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Night-time; Test type: Superiority; p = 0.6895, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.04, 95% CI 2-sided [-0.18 to 0.27], Standard Error of Mean 0.11 — (T+S_PE) - (T18GEL+S-DPI)
Statistical Analysis 7: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); Over 24 hours; Test type: Superiority; p = 0.0013, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.52, 95% CI 2-sided [-0.84 to -0.21], Standard Error of Mean 0.16 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 8: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Over 24 hours; Test type: Superiority; p = 0.0040, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.47, 95% CI 2-sided [-0.78 to -0.15], Standard Error of Mean 0.16 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 9: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Over 24 hours; Test type: Superiority; p = 0.3287, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.16, 95% CI 2-sided [-0.16 to 0.48], Standard Error of Mean 0.16 — (T+S_PE) - (T18GEL+S-DPI)

23. Secondary Outcome: Response in Mean Number of Days With Night-time Awakenings
Description: Response in mean number of days with night-time awakenings. Per treatment period, the mean number days with awakening during the night was calculated. Per 6-week treatment period the data obtained after the first 3 weeks was used for calculating this mean. Mean number of days with night-time awakenings response is defined as the change from baseline. The baseline value, mean number of days with night-time awakenings (Baseline), is defined as the mean of the number of days with night-time awakenings obtained from the last week preceding the randomization visit.
Time Frame: At baseline and last 3 weeks of 6-week treatment period.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 127 | 124 | 125
Days | -0.06 (0.03) | -0.06 (0.03) | -0.05 (0.03) | 0.07 (0.03)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.9956, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.00, 95% CI 2-sided [-0.03 to 0.03], Standard Error of Mean 0.01 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p = 0.7100, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.01, 95% CI 2-sided [-0.03 to 0.02], Standard Error of Mean 0.01 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.3659, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.01, 95% CI 2-sided [-0.02 to 0.04], Standard Error of Mean 0.01 — (T+S_PE) - (T18GEL+S-DPI)

24. Secondary Outcome: Response in Mean Number of Days With Night-time Awakenings Due to Shortness of Breath (SOB)
Description: Per treatment period, the mean number days with awakening (only chronic obstructive pulmonary disease (COPD) related awakenings) during the night was calculated. Per 6-week treatment period the data obtained after the first 3 weeks was used for calculating the mean.
  Mean number of days with COPD related awakenings response is defined as the change from baseline.
  The baseline value, mean number of days with COPD related awakenings (Baseline), is defined as the mean of the number of days with COPD related awakenings obtained from the last week preceding the randomization visit.
Time Frame: At baseline and last 3 weeks of 6-week treatment period.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 127 | 124 | 125
Days | -0.05 (0.02) | -0.04 (0.02) | -0.04 (0.02) | -0.07 (0.02)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.4416, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.01, 95% CI 2-sided [-0.04 to 0.02], Standard Error of Mean 0.01 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p = 0.7058, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.01, 95% CI 2-sided [-0.03 to 0.02], Standard Error of Mean 0.01 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.1494, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.02, 95% CI 2-sided [-0.01 to 0.05], Standard Error of Mean 0.01 — (T+S_PE) - (T18GEL+S-DPI)

25. Secondary Outcome: Response in Means Number of Awakenings Due to Shortness of Breath (SOB)
Description: Per treatment period, the mean number of awakening (only chronic obstructive pulmonary disease (COPD) related awakenings) during the night was calculated. Per 6-week treatment period the data obtained after the first 3 weeks was used for calculating this mean. Mean number of COPD related awakenings response is defined as the change from baseline. The baseline value, mean number of COPD related awakenings (Baseline), is defined as the mean of the number of days with COPD related awakenings obtained from the last week preceding the randomization visit.
Time Frame: At baseline and last 3 weeks of 6-week treatment period.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Awakenings
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 127 | 124 | 125
Awakenings | -0.02 (0.04) | -0.02 (0.04) | -0.04 (0.04) | -0.08 (0.04)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.9980, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.00, 95% CI 2-sided [-0.06 to 0.06], Standard Error of Mean 0.03 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p = 0.4618, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.02, 95% CI 2-sided [-0.04 to 0.08], Standard Error of Mean 0.03 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.0418, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.06, 95% CI 2-sided [0.00 to 0.12], Standard Error of Mean 0.03 — (T+S_PE) - (T18GEL+S-DPI)

26. Secondary Outcome: Response in Average Shortness of Breath (SOB) Score at Night
Description: Response in average shortness of breath (SOB) score at night. The SOB measured the shortness of breath, ranging from 1 to 5, where 1 = not at all, 2 = a little bit, 3 = somewhat, 4 = quite a bit and 5 = very much. A higher score indicates a worse outcome.
  Per 6-week treatment period the data obtained after the first 3 weeks was used for calculating the mean.
Time Frame: At baseline and last 3 weeks of 6-week treatment period.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 127 | 124 | 125
Score on a scale | -0.06 (0.05) | -0.04 (0.05) | -0.06 (0.05) | -0.11 (0.05)
Statistical Analysis 1: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium (Tio18GEL); Test type: Superiority; p = 0.4206, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = -0.02, 95% CI 2-sided [-0.08 to 0.03], Standard Error of Mean 0.03 — (T+S_PE) - (Tio18GEL)
Statistical Analysis 2: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 50 µg Salmeterol MDPI (Salm50DPI); Test type: Superiority; p = 0.8723, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.00, 95% CI 2-sided [-0.05 to 0.06], Standard Error of Mean 0.03 — (T+S_PE) - (Salm50DPI)
Statistical Analysis 3: Comparison: 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) vs 18 µg Tiotropium Free Combination (T18GEL+S_DPI); Test type: Superiority; p = 0.1005, ANOVA; Analysis of variance with terms for centre, patient within centre, treatment, and period. α = 0.05 two-sided; Difference of adjusted means = 0.05, 95% CI 2-sided [-0.01 to 0.11], Standard Error of Mean 0.03 — (T+S_PE) - (T18GEL+S-DPI)

27. Secondary Outcome: Number of Participants With Drug Related Adverse Events
Description: Number of participants with drug related adverse events.
Time Frame: From first drug administration until last drug administration (average duration of 42 days) + 30 days, up to 91 days for T+S_PE, up to 98 days for Tio18GEL, up 89 days for Salm50DPI and up to 113 days for T18GEL+S_DPI.
Population: Treated Set (TS): All randomised patients who took at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 132 | 135 | 137 | 132
Participants | 0 | 2 | 2 | 2

28. Secondary Outcome: Number of Patients With Marked Changes in Vital Signs
Description: Marked changes from baseline in vital signs were defined as followed:
  Systolic blood pressure
  * Increase of ≥25 millimetre of mercury (mmHg) above baseline
  * Decrease below 100 mmHg if not at that level at baseline and a decrease of >10 mmHg below baseline
  Diastolic blood pressure
  * Increase above 90 mmHg and an increase of >10 mmHg above baseline
  * Decrease below 60 mmHg if not at that level at baseline and a decrease of >10 mmHg below baseline
  Pulse
  * Increase above 100 bpm if not at that level at baseline and an increase of >10 bpm above baseline
  * Decrease below 60 bpm if not at that level at baseline and a decrease of >10 bpm below baseline
  Baseline is defined as the pre-dose measurement at randomisation visit.
Time Frame: At baseline and 6 hours following the morning dose of study medication after 6 weeks of treatment.
Population: Treated Set (TS): All randomised patients who took at least one dose of study medication and who had available data.
Measure: Count of Participants; unit: Participants
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI)
Number analyzed (Participants) | 127 | 128 | 125 | 127
Participants
  Increase in systolic blood pressure | 18 | 18 | 16 | 15
  Increase in diastolic blood pressure | 16 | 16 | 11 | 14
  Increase in pulse rate | 6 | 10 | 9 | 13
  Decrease in systolic blood pressure | 3 | 4 | 3 | 4
  Decrease in diastolic blood pressure | 5 | 7 | 3 | 5
  Decrease in pulse rate | 6 | 7 | 7 | 2

ADVERSE EVENTS:
Time Frame: From first drug administration until last drug administration (average duration of 42 days) + 30 days, up to 91 days for T+S_PE, up to 98 days for Tio18GEL, up 89 days for Salm50DPI and up to 113 days for T18GEL+S_DPI.
Description: Treated Set (TS): All randomised patients who took at least one dose of study medication.
Groups:
- Total Treated: All patients who received at least one dose of study medication.
Arm/Group | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) | 18 µg Tiotropium (Tio18GEL) | 50 µg Salmeterol MDPI (Salm50DPI) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI) | Total Treated
All-Cause Mortality (participants affected / at risk) | 0/132 | 1/135 | 0/137 | 0/132 | 1/146
Serious Adverse Events (participants affected / at risk) | 1/132 | 7/135 | 4/137 | 2/132 | 13/146
Other Adverse Events (participants affected / at risk) | 14/132 | 15/135 | 14/137 | 11/132 | 47/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) (N=132) | 18 µg Tiotropium (Tio18GEL) (N=135) | 50 µg Salmeterol MDPI (Salm50DPI) (N=137) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI) (N=132) | Total Treated (N=146)
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 0 | 3
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Meningitis pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 7.5 µg /25 µg Tio /Salmeterol (T+S_PE) (N=132) | 18 µg Tiotropium (Tio18GEL) (N=135) | 50 µg Salmeterol MDPI (Salm50DPI) (N=137) | 18 µg Tiotropium Free Combination (T18GEL+S_DPI) (N=132) | Total Treated (N=146)
Nasopharyngitis (Infections and infestations) | 9 | 9 | 7 | 6 | 27
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 7 | 3 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.